CLINICAL TRIAL: NCT05540041
Title: The Efficacy of Bubble Breathing Play Therapy and Tell-show-do Play Therapy in the Preoperative Anxiety Children and Their Parent
Brief Title: Reducing Anxiety of Children and Their Parents in the Pre-Operative Process With Therapeutic Play
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Isparta University of Applied Sciences (Other)
Collaborators: Akdeniz University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IspartaUAS3
Record Dates: First submitted 2022-09-09; First posted 2022-09-14 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Preoperative Care; Child; Parents; Anxiety
Keywords: Preoperative Care; Child; Parents; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Masking Description: Single (Participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bubble breathing play therapy (Experimental): Children in intervention group 2 will be given a bubble breathing play therapy intervention. With this intervention, it is aimed to teach the child and parent to breathe correctly and deeply, to relax them, to reduce their anxiety and fears, to relax, to direct their attention to something other than pain. In the intervention pediatric surgery service, investigative coaching will be applied 30 minutes before premedication. The procedure time is planned to be at least 5-10 minutes. The intervention will be implemented with a ready-made foam bubble toy. The toy will be provided by the researcher and given to the children as a gift.
  Interventions: Other: Bubble breathing play therapy group
- Tell-show-do play therapy (Experimental): Tell-show-do play therapy initiative will be applied to children included in intervention group 1. The initiative will be applied to children without disturbing the parent-child relationship. The intervention will be applied for 10-15 minutes. The tell-show-do play therapy initiative will be implemented using the directed play therapy method and therapeutic play tools. Amigurumi dolls, medical toys (surgical shirt, movable toy bed) and real medical materials such as stethoscope, patient armband, bone, mask, degree will be used as therapeutic play tools.
  Interventions: Other: Tell-show-do play therapy group
- No intervention (Other): The participants in the control group will be given routine nursing care.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: Bubble breathing play therapy group — The efficacy of bubble breathing play therapy in the preoperative anxiety children and their parent.
  Arms: Bubble breathing play therapy
Other: Tell-show-do play therapy group — The efficacy of tell-show-do play therapy in the preoperative anxiety children and their parent.
  Arms: Tell-show-do play therapy
Other: No intervention — Routine nursing care
  Arms: No intervention

SUMMARY:
It is emphasized in studies that child and parent anxiety that arises in pediatric surgery should be prevented or reduced. According to previous studies, one way to reduce child and parent anxiety in the preoperative period is therapeutic play interventions. This study was planned to compare the effectiveness of two different therapeutic play interventions (bubble breathing play therapy and tell-show-do play therapy) in reducing preoperative anxiety of children and parents who are scheduled for elective surgery.

DETAILED DESCRIPTION:
Aim: This study was planned to comparison of the effectiveness of two different therapeutic play interventions (bubble breathing play therapy and tell-show-do play therapy) in reducing preoperative anxiety of children and parents who are scheduled for elective surgery.

Method: This study was planned as a randomized controlled trial. The sample of the study will consist of 105 children aged 5-12, who will be operated on at Akdeniz University Hospital, and their parents. Randomization result; It was planned to include a total of 105 children and their parents in 3 groups: bubble breathing play therapy group (intervention group 1)= 35, tell-show-do play therapy group (intervention group 2)= 35 , and control group= 35 children and parents.

Child and parent information form will be used to collect data, Modified Yale Preoperative Anxiety Scale will be used to collect data in child sample, and Spielberger State Anxiety Scale will be used to collect data in parent sample.

Intervention and Data Collection: Randomization will be performed after the purpose of the study is explained to the child and parent who agreed to participate in the study and after obtaining consent. Immediately after the pretest (first measurement) is given to the children assigned to intervention group 1 and their parents, attempts to bubble breathing play therapy will be applied for 5-10 minutes. If they wish, the child and parents will be told that they can continue to play with the bubble toys until premedication. Children assigned to intervention group 2 and their parents will be tell-show-do play therapy for 10-15 minutes immediately after the pre-test (first measurement) is done. Participants randomized to the control group will be given routine standard nursing care. The second measurement will be just before premedication (post test). Thus, the effectiveness of the initiatives and their comparison with each other will be evaluated.

The data of the research will be analyzed using the Statistical Package of Social Science (SPSS) 23.0 software package program. The process of evaluating the data will be carried out with the support of a statistician.

ELIGIBILITY:
Inclusion Criteria:

* Being a child between the ages of 5-12 for which a surgical operation is planned
* Being the parent of a child between the ages of 5 and 12 whose surgical operation is planned
* Not having vision, hearing or speech problems
* Not have a mental or neurological disability
* Not being diagnosed with an anxiety disorder
* Children and parents who can speak and understand Turkish will be included in the study

Exclusion Criteria:

* Change in surgical operation date
* Using another distraction technique

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 210 (Estimated)
Dates: Start 2022-10-18 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Preoperative anxiety of children | Anxiety levels of children will be evaluated twice. The first measurement will be made 30 minutes before the premedication, and the last measurement will be made just before the premedication.
  The decrease in anxiety levels of children whose attention is diverted with play dough and kaleidoscope is an outcome measure. This decrease will be measured with the "Modified Yale Preoperative Anxiety Scale". Outcome criteria will be evaluated twice in Pediatric Surgery Service, approximately 30 minutes before premedication and just before premedication (pretest-posttest). The scale consists of twenty-two items and five categories. Each category gets one point out of four. The higher the score on the scale, the greater anxiety. In the post-test, it will be evaluated whether there is a decrease according to the pre-test score. If there is a decrease in the "posttest" scores compared to the "pretest" scores, it can be said that distraction positively affects preoperative anxiety. Statistical significance will be set to p < 0.05.
Preoperative anxiety of parent | Anxiety levels of parents will be evaluated twice. The first measurement will be made 30 minutes before the premedication, and the last measurement will be made just before the premedication.
  The decrease in anxiety levels of parents of children whose attention is diverted with play dough and kaleidoscope is an outcome measure. This decrease will be measured by the "Spielberger State Anxiety Scale". Outcome criteria will be evaluated twice in Pediatric Surgery Service, approximately 30 minutes before premedication and just before premedication (pretest-posttest). The 4-point Likert-type scale, consisting of 20 items in total, measures the anxiety of the person at a certain time. For scores above 42 points, it indicates a high level of anxiety. In the post-test, it will be evaluated whether there is a decrease according to the pre-test score. If there is a decrease in the "posttest" scores compared to the "pretest" scores, it can be said that distraction positively affects preoperative anxiety. Statistical significance will be set to p < 0.05.

CONTACTS AND LOCATIONS:
Overall Officials: Fahriye RN PAZARCIKCI, PhD, Study Director — Isparta University of Applied Sciences; Emine RN EFE, Professor, Study Chair — Akdeniz University; Şevkiye DİKMEN, Study Chair — Akdeniz University; Öznur ARAYAN, Study Chair — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Antalya/Merkez, Turkey (Türkiye)

REFERENCES:
- [Background] Azher U, Srinath SK, Nayak M. Effectiveness of Bubble Breath Play Therapy in the Dental Management of Anxious Children: A Pilot Study. J Contemp Dent Pract. 2020 Jan 1;21(1):17-21. PMID 32381795
- [Background] Sridhar S, Suprabha BS, Shenoy R, Shwetha KT, Rao A. Effect of a relaxation training exercise on behaviour, anxiety, and pain during buccal infiltration anaesthesia in children: Randomized clinical trial. Int J Paediatr Dent. 2019 Sep;29(5):596-602. doi: 10.1111/ipd.12497. Epub 2019 Apr 8. PMID 30887592